CLINICAL TRIAL: NCT04193462
Title: A Brief Relationship-Based Intervention for Post-Partum Depression; Effects on Mother's Hormones, Depression and Parenting and on Infant Social-Emotional Development
Brief Title: Relationship-Based Intervention for Post-Partum Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Interdisciplinary Center Herzliya (Other)
Responsible Party: Principal Investigator, Moran Influs, Principal Investigator, Interdisciplinary Center Herzliya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: InterdisciplinaryCH
Record Dates: First submitted 2019-11-01; First posted 2019-12-10 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Post Partum Depression
Keywords: Post-partum depression; dyadic psychotherapy; oxytocin
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Post-partum depression- Dyadic psychotherapy (Experimental): Mothers and infants will be treated with 8 weeks dyadic psychotherapy at their home using video-feedback of mother-infant interaction to discuss main issues in the mother-infant relationship.
  Interventions: Other: Post-partum depression- Dyadic psychotherapy-
- Post-partum depression- Psycho-educational therapy (Active Comparator): 8 weeks of supportive therapy for the mother at her house, involving the baby. Each session will include different aspects of psycho-education regarding development of the baby.
  Interventions: Other: Post-partum depression- Psycho-educational therapy
- Control- Healthy mothers and their babies (No Intervention): No intervention for 8 weeks.

INTERVENTIONS:
Other: Post-partum depression- Dyadic psychotherapy- — Mothers and infants will be treated with dyadic psychotherapy focused on interactions, emphasizing eye contact, body language, empathy, and social reciprocity. Dyadic psychotherapy will be administered one time a week during the 8-week trial period, at the subject's home. Each session, approximately 90 minutes long, will include videotaping mother-infant interaction, watching the last session's interaction as a part of video-feedback technique, and discussing main issues in the mother-infant relationship. In addition, each session will begin and end with a- 5-minute episode of affectionate touch and gaze synchrony between the mother and her infant. During the whole therapy-trial, the therapist will also use cognitive-behavioral approach to address the mother's perception of her infant and of herself as a mother.
  Arms: Post-partum depression- Dyadic psychotherapy
Other: Post-partum depression- Psycho-educational therapy — Mothers will receive a therapy in their homes for 8 weeks, 1.5 hours for each session by a therapist arriving at their home. Each session will address a different developmental aspects of the baby (feeding, movement, social-emotional development etc.). Therapist will ask the mother about her baby, will give information about developmental needs and expectations and will help mother to enrich child's development and deal will potential problems
  Arms: Post-partum depression- Psycho-educational therapy

SUMMARY:
A short term dyadic psychotherapy intervention for mothers with Post-Partum depression and their babies in the first year of life was developed. The investigators believe that following dyadic intervention mothers will show improvement in depressive symptoms, the quality of the mother-child relationship will improve, and maternal and infant's oxytocin levels will rise.

DETAILED DESCRIPTION:
Subjects: 60 Mothers will be interviewed and diagnosed as suffering from Post-Partum- depression (PPD) according to the Diagnostic and Statistical Manual of Mental Disorders, IV version (DSM-IV), enrolling within 3-8 months postpartum. Mothers will be recruited through social media networks. Additional 40 mothers, 3-8 months postpartum will be assessed and diagnosed as not suffering from PPD or any other psychiatric psychopathology.

Procedure: The baseline assessment will be conducted at the infant's home. A parent-infant interaction will be videotaped and salivary oxytocin samples will be collected from the infant and from the mother.

The women in the PPD group will participate in 8 weeks of dyadic psychotherapy (DP) combining video feedback, or a psycho-educational treatment regarding child development (randomize selection will be made). During the 8-week treatment, salivary oxytocin samples will be collected from the infants and from the mother at the beginning and the end of each session.

Another assessment will be conducted at the infant's home, at the end of the treatment. As in the baseline condition, this assessment will include videotaped parent-infant interaction, as well as salivary oxytocin samples collection from the mother and from the infant. Parent-infant interaction will be filmed and assessed using the CIB Manual (Feldman, 1998) and the synchrony coding system.

Healthy mothers will undergo the same baseline assessment and a second assessment within 2-3 months, and won't get any treatment.

ELIGIBILITY:
Inclusion Criteria:

* women diagnosed with Post-Partum depression, major or minor, according to the Diagnostic and Statistical Manual of Mental Disorders, 5th version (DSM-5)
* 3-8 months after birth of one baby

Exclusion Criteria:

* Mothers of twins
* Mothers of premature babies
* Comorbidity of psychopathology, women who have severe personality disorder or other psychiatric diagnose, besides depression or anxiety
* Women or babies who suffer from severe medical condition, such as developmental problems for the baby or disability.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Behavioral Assessment of dialogue | trail 1-baseline
  Interactions will be coded with the "Coding Interactive Behavior" (CIB) manual (Feldman, 1998), infant version. This version is composed of 37 codes rated on a scale of 1 to 5, as higher score means a better outcome.
Hormonal Assays- Oxytocin | trail 1-baseline
  Three saliva samples will be collected using Salivettes® at baseline, following interaction, and 20 minutes after end and averaged. All samples will be then stored at -20°C. Salivette will be treated as following: centrifuged twice, at 4°C at 1500 x g for 30 minutes, aliquoted and lyophilized over few days- to concentrate by 4 times. The dry samples will be reconstructed in the assay buffer immediately before analysis using an oxytocin enzyme immunoassay commercial kit (ENZO, NY). The assay preformed according the kit's instruction. The concentration of oxytocin will be calculated using MatLab-7

SECONDARY OUTCOMES:
Behavioral Assessment of dialogue | trail 2- after treatment- 2-3 months after trail 1
  Interactions will be coded with the "Coding Interactive Behavior" (CIB) manual (Feldman, 1998), infant version. This version is composed of 37 codes rated on a scale of 1 to 5, as higher score means a better outcome.
Hormonal Assays- Oxytocin | trail 2- after treatment- 2-3 months after trail 1
  Three saliva samples will be collected using Salivettes® at baseline, following interaction, and 20 minutes after end and averaged. All samples will be then stored at -20°C. Salivette will be treated as following: centrifuged twice, at 4°C at 1500 x g for 30 minutes, aliquoted and lyophilized over few days- to concentrate by 4 times. The dry samples will be reconstructed in the assay buffer immediately before analysis using an oxytocin enzyme immunoassay commercial kit (ENZO, NY). The assay preformed according the kit's instruction. The concentration of oxytocin will be calculated using MatLab-7

CONTACTS AND LOCATIONS:
Overall Officials: Moran Influs, Phd, Study Director — Interdisciplinary Center Herzliya, Israel
Locations (1):
- Interdisciplinary Center, Herzliya, Israel